CLINICAL TRIAL: NCT05611489
Title: Laparoscopic Versus Open Appendectomy Prospective Randomized Control Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abanoub Atif Fawzy (Other)
Responsible Party: Sponsor-Investigator, Abanoub Atif Fawzy, Principle investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laparoscopic appendectomy
Record Dates: First submitted 2022-11-01; First posted 2022-11-10 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Appendicitis Acute
Keywords: Laparoscopic appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: laparoscopic versus open appendectomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open appendectomy (Other): Appendectomy will be done through Mcberney incision.
  Interventions: Procedure: Open appendectomy
- Conventional lap appendectomy (Other): Three ports will be inserted as follows: One 10/12 umbilical port, one 5mm suprapubic (or right suprapubic)port, one 5mm or 10/12mm port in left iliac fossa (or left suprapubic).
  Interventions: Procedure: Conventional Lap appendectomy

INTERVENTIONS:
Procedure: Open appendectomy — performed With the patient in supine position.incision made lateral to McBurney's point.layers of the abdomen is exposed. If the cecum can be visualized, it can be mobilized and used to identify the appendix. Once the appendix is identified, the mesoappendix should be dissected and the appendiceal vessels divided between clamps. The appendiceal vessels are then ligated with silk sutures. A silk purse-string suture can then be placed around the appendiceal base.A 15-blade knife is then used to excise the appendix proximal to the right angle clamp.The appendiceal stump mucosa can be obliterated using electrocautery. Then good haemostasis and layered closure is done.
  Arms: Open appendectomy
Procedure: Conventional Lap appendectomy — Three ports will be inserted as follows: One 10/12 umbilical port, one 5mm suprapubic (or right suprapubic)port, one 5mm or 10/12mm port in left iliac fossa (or left suprapubic). One additional trocar can be inserted following surgeons preference. Retraction of the appendix would be performed with a forceps. The mesoappendix will be divided with bipolar or monopolar cautery. The appendix stump will be ligated with suture loop or with an endo-stapler. The specimen will be delivered within a plastic bag or in any protected way (without any contact with the abdominal wall) via the umbilical port. Any fluid will be suctioned and washing performed if required. Fascial defects (10/12 trocars)will be closed with 2-O polydioxanone sutures and skin closed with 4-O non-absorbable sutures. No pelvic drain will be inserted. A three-band dressing will be applied in the end.
  Other Names: Multiport Lap appendectomy
  Arms: Conventional lap appendectomy

SUMMARY:
laparoscopic versus open appendectomy prospective randomized control study.Both surgical methods are safe and well established in clinical practice but there has been a controversy about which surgical procedure is the most appropriate in this research we are going to demonstrate which operative procedure is more beneficial with less disadvantages.

DETAILED DESCRIPTION:
A double-blind study is one in which neither the participants nor the experimenters know who is receiving a particular treatment. This procedure is utilized to prevent bias in research results. Using envelopes as an allocation concealment method. Each patient will receive two envelopes one contain paper which determine that patient will have open surgery and the other determine that patient will have lap surgery and neither patient nor experimenters know about them and patient shall choose one of them which will determine what surgery will patient undergo .

ELIGIBILITY:
Inclusion Criteria:

1. patient age between 5-50 year old
2. patient diagnosed as acute appendicitis

Exclusion Criteria:

1. pregnacy
2. perforated appendix
3. severe obese patient
4. previous abdominal exploration

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Operative time | 1 year
  Time needed for operation

IPD SHARING:
Plan to Share IPD: No